CLINICAL TRIAL: NCT00431678
Title: A Multinational, Prospective, Randomized, Double-blind Study to Investigate the Efficacy and Safety of Sequential Intravenous/Oral Moxifloxacin in Comparison to Intravenous Levofloxacin Plus Intravenous Ceftriaxone Followed by Oral Levofloxacin, in the Treatment of Patients With Severe Community-acquired Pneumonia
Brief Title: Efficacy and Safety of Sequential IV/PO Moxifloxacin in Comparison to IV Levofloxacin Plus IV Ceftriaxone Followed by PO Levofloxacin, in the Treatment of Patients With Community-acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11215
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Pneumonia
Keywords: Community-acquired Pneumonia
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Moxifloxacin; Levofloxacin; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)
- Arm 2 (Active Comparator)
  Interventions: Drug: Levofloxacin + Ceftriaxone

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Sequential intravenous/oral (400/400 mg once daily for 7 to 14 days) of Avelox (Moxifloxacin, BAY12-8039)
  Arms: Arm 1
Drug: Levofloxacin + Ceftriaxone — Intravenous combination therapy of levofloxacin 500 mg twice daily and ceftriaxone (2 g once a day) followed by oral levofloxacin (500 mg twice a day for 7 to 14 days).
  Arms: Arm 2

SUMMARY:
Sequential therapy with intravenous to oral moxifloxacin, was tested at 69 study centres in 17 countries to determine if this treatment regimen is safe and effective in treating hospitalized adult patients with community-acquired pneumonia. 748 patients were participated in the study over an 18 months period. Individual patient involvement in the study was approximately 4-6 weeks. Moxifloxacin was compared to a combination treatment regimen of high dose intravenous ceftriaxone plus high dose intravenous levofloxacin followed by high dose oral levofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* All of the following signs and symptoms of pneumonia:

  * Fever (core/ rectal/ tympanic temperature >/= 38.5°C or axillary/ oral/ cutaneous temperature >/= 38.0°C) or hypothermia (core/ rectal/ tympanic temperature </= 35.5°C or axillary/ oral/ cutaneous temperature </= 35.0°C)
  * White blood cell (WBC) count > 10,000/µL, or >/= 15% immature neutrophils (bands), regardless of the peripheral WBC count, or total WBC count < 4,500/µL
  * The presence of at least 2 of the following symptoms: - Cough- Purulent sputum production
* Dyspnoea or tachypnoea (respiratory rate > 20 breaths/minute)
* Rigors and/or chills- Chest pain
* Auscultatory findings on pulmonary examination of rales/crackles and/or evidence of pulmonary consolidationAND
* Radiological evidence of (an) infiltrate(s) consistent with bacterial pneumonia at baseline or within 24 hours following enrolment
* Fine score >/= 71 (i.e. Pneumonia PSI risk Class III, IV or V, requiring hospitalisation for the treatment of CAP)
* Written informed consent obtained from the patient or a next-of-kin

Exclusion Criteria:

* Known hypersensitivity to fluoroquinolones, or other quinolones, and/or to beta-lactams, or any of the excipients
* Female patients who are pregnant or lactating
* History of tendon disease/disorder related to quinolone treatment
* Known congenital or documented-acquired QT prolongation; concomitant use of drugs, reported to increase the QT interval; uncorrected hypokalaemia; clinically relevant bradycardia; clinically relevant heart failure with reduced left
* ventricular ejection fraction; previous history of symptomatic arrhythmias
* History of epilepsy- Known glucose-6-phosphate dehydrogenase deficiency
* Known severe impaired liver function (i.e. Child Pugh C), (refer to Section 10.4 for definition) or transaminases increase > 5 fold ULN- Hospitalisation for > 48 hours before developing pneumonia, or discharge from hospital < 30 days prior- Systemic antibacterial therapy for more than 24 hours within 14 days of enrolment
* Patients requiring concomitant systemic antibacterial agents
* Known structural lung disease (e.g. cystic fibrosis, bronchiectasis, or lung cancer), or other known conditions (e.g. malnutrition) predisposing to infection with nosocomial-like organisms such as Pseudomonas aeruginosa
* Lung abscess, pleural empyema, risk factors for aspiration pneumonia (e.g. recent stroke, head injury, dementia)
* Known rapidly fatal underlying disease (death expected within 6 months)
* Known or suspected active tuberculosis or endemic fungal infection- Neutropenia (neutrophil count < 1,000/µL) caused by immunosuppressive therapy or malignancy
* Patients known to have AIDS (CD4 count < 200/µL) or HIV-seropositive patients receiving HAART
* Previous enrolment in this study
* Participation in any clinical investigational drug study within the previous 4 weeks
* Patient with pre-terminal renal failure (creatinine clearance < 10 mL/min) and patients undergoing haemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2004-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Clinical response | 5 to 7 days after last dose of study medication

SECONDARY OUTCOMES:
Clinical and bacteriological response | At the day of switch from intravenous to oral therapy
Clinical and bacteriological response on treatment | At day 3 to 5
Clinical and bacteriological response | At the end of treatment
Bacteriological response | 5-7 days after end of treatment
Mortality attributable to pneumonia | 5-7 days after end of treatment
Clinical and bacteriological response | At days 21 to 28 after end of treatment
Symptoms course of community-acquired pneumonia | at defined visits
Adverse Event Collection | all visits

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (82):
- Argentina (2):
  - Vicente López, Buenos Aires
  - Buenos Aires, Buenos Aires F.D.
- Belgium (4):
  - Bruxelles - Brussel
  - Leuven
  - Liège
  - Namur
- Chile (3):
  - Temuco, Región de la Araucanía
  - Viña del Mar, Región de Valparaíso
  - Santiago
- Colombia (2):
  - Bogotá
  - Bucaramanga
- France (11):
  - Agen
  - Aix-en-Provence
  - Argenteuil
  - Avignon
  - Belfort
  - Bordeaux
  - Brive-la-Gaillarde
  - Paris
  - Saint-Gaudens
  - Toulon
  - Vesoul
- Germany (6):
  - Bochum, North Rhine-Westphalia
  - Lüdenscheid, North Rhine-Westphalia
  - Paderborn, North Rhine-Westphalia
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Greece (3):
  - Rio, Patras
  - Thessaloniki, Thessaloniki
  - Athens
- Israel (5):
  - Afula, Israel
  - Ashkelon, Israel
  - Holon, Israel
  - Tel Aviv, Israel
  - Tel Litwinsky
- Lithuania (2):
  - Kaunas
  - Vilnius
- Mexico (4):
  - Toluca, Edo. de México
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - México, D.F.
- Netherlands (5):
  - Eindhoven, North Brabant
  - 's-Hertogenbosch
  - Ede
  - Harderwijk
  - Heerlen
- Peru (3):
  - Callao
  - Lima
  - Lima Cercado
- Poland (6):
  - Bydgoszcz
  - Gdansk
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw
- Lisbon, Portugal
- South Africa (7):
  - Bloemfontein, Free State
  - Bloemfontein, Freestate
  - Brits, Gauteng
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Cape Town, Western Cape
  - Somerset West, Western Cape
- Spain (7):
  - Huesca, Aragon
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Guadalajara, Guadalajara
  - Alcalá de Henares, Madrid
  - Madrid, Madrid
  - Valencia, Valencia
- Sweden (4):
  - Jönköping
  - Kalmar
  - Karlstad
  - Skövde
- United Kingdom (7):
  - Middlesbrough, Cleveland
  - Dumfries, Dumfries and Galloway
  - Hull, Humberside
  - Edinburgh, Lothian
  - Rotherham, South Yorkshire
  - Sheffield, South Yorkshire
  - Newcastle upon Tyne, Tyne and Wear

REFERENCES:
- [Derived] Torres A, Garau J, Arvis P, Carlet J, Choudhri S, Kureishi A, Le Berre MA, Lode H, Winter J, Read RC; MOTIV (MOxifloxacin Treatment IV) Study Group. Moxifloxacin monotherapy is effective in hospitalized patients with community-acquired pneumonia: the MOTIV study--a randomized clinical trial. Clin Infect Dis. 2008 May 15;46(10):1499-509. doi: 10.1086/587519. PMID 18419482